CLINICAL TRIAL: NCT06035913
Title: Doctor of Medicine, Chief Physician, Associate Professor, Master Supervisor, Administrative Deputy Director of Neurology.
Brief Title: Mid-and Long-term Efficacy of Ergot Alkaloids in the Treatment of Salivation in Patients With Parkinson's Disease.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20230829-01
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Main Heading (Descriptor) Terms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Salivation group: The saliva group was instructed to take dihydroergot mesylate, one tablet twice a day, and observed the improvement of salivation after 1 week, after 1 month, after March and after 6 months.
  Interventions: Drug: Dihydroergot mesylate

INTERVENTIONS:
Drug: Dihydroergot mesylate — take medicine

SUMMARY:
Parkinson's disease is the second most common neurodegenerative disease after Alzheimer's disease, the incidence of population over 60 years old in China is 1.37%, Parkinson's disease is often accompanied by various non-motor symptoms, such as salivation. Salivation can occur at any time in Parkinson's disease, with an incidence of 32% to 74%, often leading to social embarrassment, skin infections, bad breath, aspiration pneumonia, etc. This not only reduces the quality of life of patients, but also increases the burden on caregivers. Salivation can improve symptoms with botulinum toxin injections, medications, and non-drug treatments. Dihydroergot mesylate has been shown to be effective in the treatment of salivation in patients with Parkinson's disease, and this study will further observe the medium- to long-term efficacy of the drug on salivation symptoms.

DETAILED DESCRIPTION:
The objective of the study is to further observe the medium- and long-term efficacy and adverse reactions of the drug on the basis of the proven effectiveness of dihydroergot mesylate sustained-release tablets on salivation symptoms in patients with Parkinson's disease, and to evaluate the effect of the drug on swallowing function and cognitive function of patients and explore its possible mechanism of action. The study was based on a scale assessment of identified cases, and at the identified endpoints, the primary outcome was set as improvement in SCS-PD scale scores after March, and secondary outcomes were set as disease progression since March (as demonstrated by MDS-UPDRS Part III scale scores), changes in swallowing function, cognitive function, liver and kidney function indicators, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

Age: Adult (≥ 18 years) Gender: male or female All patients met the British Parkinson's Association Brain Bank criteria for the clinical diagnosis of primary Parkinson's disease Patients had mild, moderate, to severe salivation (MDS-UPDRS-IL-2 score≥ 2) There has been no drug adjustment in the past 3 months Voluntarily sign an informed consent form

Exclusion Criteria:

Secondary PD or Parkinson's superposition syndrome Those with severe cognitive impairment, speech impairment, dysarthria, and deafness who cannot cooperate with the completion of the examination History of previous drug allergy Have a condition other than Parkinson's disease that can cause severe salivation or other oral and glandular problems In the past 3 months, botulinum toxin, anticholinergic drugs, etc. have been used to treat salivation symptoms Severe cardiopulmonary diseases, tumors, liver and kidney diseases and other chronic wasting diseases People with mental disorders No previous history of dysphagia or salivation due to cerebral infarction or other causes Those who do not cooperate with the test requirements process and follow-up Those who had poor medication adherence during the study, including alcohol abuse and drug dependence Subjects enrolled in clinical trials of other drugs within 3 months Severe orthostatic hypotension and bradycardia and organic lesions of the heart, decreased renal function Subjects who the investigators consider unsuitable for clinical trials for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the diagnostic criteria for Parkinson's disease and have varying degrees of salivation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of the SCS-PD scale | 6 months
  Improvement in salivation was assessed by the change in scores on the SCS-PD scale

CONTACTS AND LOCATIONS:
Overall Officials: Youyong Tian, Study Director — Chief physician
Locations (1):
- Dihydroergot mesylate, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No